CLINICAL TRIAL: NCT00173199
Title: The Changes of Cytokines in Guillain Barré Syndrome: the Correlation With Clinical Manifestations and Skin Innervation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700526
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-06

CONDITIONS: Guillain Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
In order to increase our understanding about the pathogenic mechanism and the strategy of treatment in the subtypes of Guillain Barré syndrome, we will check the temporal changes of cytokines with different biological activities in serum and cerebrospinal fluid (CSF), check the titer of various anti-ganglioside antibodies, perform skin biopsy and correlate these data with the clinical findings such as severity and prognosis

DETAILED DESCRIPTION:
In the past the nerve system has long been regarded as a privileged site of immune system due to (1) the absence of lymphatic drainage, which limits the immunological circulation; (2) the blood-brain barrier (BBB) or blood-nerve barrier (BNB), which limits the passage of immune cells and factors; (3) the low level of expression of MHC factors, particularly MHC II, in the resident cells of the nerve system and the lack of potent antigen presenting cells, such as dendritic or Langerhans' cells, both of which lead to reduced recognition of the neurons or nerves by the immune system; and (4) the presence of immunosuppressive factors such as TGF-b. which suppress the immune response in the nervous system.

However in the past few years, the concept of privilege is revised, that is the differences in the immunological aspects between the nervous system and other organs are more quantitative than absolutely qualitative. Several lines of evidence indicate that BBB and BNB are not complete both anatomically and functionally and activated T cells can cross these barriers and traffic in and out the nervous system. The nervous system also contains a collection of immunologically resident cells, including professional or non-professional antigen presenting cells such as resident endoneurial or perivascular macrophage, glial cells, Schwann cells and endoneurial capillary endothelial cells, which are capable of synthesizing cytokines that were initially classified within the domain of the immune system and are found to express a range of appropriate specific receptors, both characteristics mediate the immunological processes in the nervous system.

The nerve system is therefore a target of immune attacks. Many disorders of the central or peripheral nerve system are related to activation of the immune system. Immune mechanisms seem important in the pathogenesis and treatments of these disorders.

Cytokines are a diverse group of soluble proteins and peptides which act as humoral regulators and modulate the activities of individual cells and tissues either under normal or pathological condition. Unlike the hormone, cytokines are usually made by more than one type of cells, have multiple target cells and multiple actions, and usually function in short acting radius. Constitutive cytokine production is usually low or absent and its production is promoted by certain stimuli at the transcription and translation level. The functions of cytokine are pleitropic and redundant. In embryogenesis and organ development, it acts as a regulator of miosis, differentiation, migration, cell growth and cell death; and in host defense response to infection, inflammation, autoimmune, trauma and metabolic injury, it not only stimulate immune cells to proliferate and differentiate but also regulate the progression and termination of immunological reaction. Some cytokines that make the inflammation progress are referred as pro-inflammatory cytokines. The major pro-inflammatory cytokines that are responsible for early responses are IL1, IL6, and TNF-alpha. Other pro-inflammatory mediators include IFN-gamma, TGF-beta, GM-CSF, IL11, IL12, IL17, IL18, IL8 and a variety of other chemokines that chemoattract inflammatory cells. When these cytokines are produced or administered into human, they induce destruction of tissues, up-regulation of the synthesis of other pro-inflammatory cytokines by various immunological cells, and induction of systemic inflammatory reaction like fever and shock. Another immunoregulatory cytokines that counteract the inflammation or the production of pro-inflammatory cytokines are referred as anti-inflammatory cytokines. These mediators act mainly by the inhibiting the production of pro-inflammatory cytokines or by counteracting many biological effects of pro-inflammatory mediators and thus contribute to the control of the inflammatory responses. The major anti-inflammatory cytokines are IL4, IL10, and IL13. Other anti-inflammatory mediators are IL16, IFN-alpha, TGF-beta, G-CSF, as well as soluble receptors for TNF or IL6. It is supposed that the balance between pro-inflammatory cytokines and anti-inflammatory cytokines determines the net effect of an inflammatory response. In addition, cytokine responses are regulated by special subpopulations of CD4 (+) T-cells, called helper T cell. They provide help to other cells of the immune system in mounting immune responses by causing cell activation or the secretion of cytokines. Th1 cells stimulate strong cellular immunity but only weak and transient antibody responses. These cells produce a number of cytokines known asTh1 cytokines and including IL2, IFN-gamma, IL12 and TNF-beta. In contrast Th2 cells evoke strong antibody responses but relatively weak cellular activity. These cells produce cytokines that are known as Th2 cytokines and include IL4, IL5, IL6, IL10, and IL13. Th1 and Th2 cells can keep each other in check and prevent inflammatory reactions in response to pathogens getting out of control. However, imbalances may also precipitate inappropriate reactions. It is thought that some autoimmune disorders and allergies may be related to overactive Th1 or Th2 responses.

Guillain-Barré syndrome (GBS) is clinically defined as an acute peripheral neuropathy over a time period of days or, at the most, up to 4 weeks. GBS may not be a single disease, but a variety of acute neuropathies with different clinical and electrophysiological manifestations. GBS is considered to be an autoimmune disease caused by cross reaction of infectious agents with auto-antigen. The triggering of autoimmunity depends both on the increase in immunogenicity of the target cell and the individual's own capability to recognize the antoantigens (HLA genes, T cell repertoire). The pathogenesis of GBS is not yet fully understood and GBS with variable clinical manifestations are supposed to be associated different immune mediated pathogenic mechanisms. By studying the GBS patients about their clinical manifestations, conventional laboratory studies, electrophysiological studies and skin biopsies and by evaluating the cytokine expression in the CSF and serum in different subtypes of GBS, we want to clarify the relationship between the immunological parameters and the clinical manifestations in GBS.

ELIGIBILITY:
Inclusion Criteria:

* Progressive weakness of both legs and arms; areflexia; cranial nerve involvement (such as facial palsies); progression over days to 4 wks; recovery beginning 2-4 wks after progression ceases; elevated cerebrospinal fluid protein with <10 cells/µl; electrodiagnostic features of nerve conduction slowing or block.

Exclusion criteria:

* nil

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, PhD, Study Director — Department of Anatomy and Cell Biology, National Taiwan University College of Medicine; Department of Neurology, National Taiwan University Hospital
Locations (1):
- Department of Anatomy and Cell Biology, National Taiwan University College of Medicine, Taipei, Taiwan